CLINICAL TRIAL: NCT03185546
Title: Project 2: The Impact of Cigarette Nicotine Content, E-cigarette Nicotine Content, and E-cigarette Flavoring on Smoking Behavior
Brief Title: Project 2 Cigarette and E-cigarette Nicotine Content and E-liquid Flavors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of Pennsylvania (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00047676; 1U54DA031659-01 (NIH); U54DA031659-06 (NIH)
Record Dates: First submitted 2017-05-22; First posted 2017-06-14 (Actual); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Smoking
Keywords: smoking; vaping
MeSH Terms: conditions — Smoking; Vaping | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Normal Nicotine Content (NNC) cigarette + moderate nicotine e-liquid + tobacco flavors (Experimental): Participants are provided with normal nicotine content tobacco Spectrum Cigarettes along with moderate nicotine level e-liquid cartridges and can choose from tobacco e-liquid flavors.
  Interventions: Other: NNC Spectrum Cigarette; Other: Moderate nicotine level e-liquid; Other: Tobacco Flavors
- NNC cigarette + low nicotine e-liquid + tobacco flavors (Experimental): Participants are provided with normal nicotine content tobacco Spectrum Cigarettes along with very low nicotine level e-liquid cartridges and can choose from tobacco e-liquid flavors.
  Interventions: Other: NNC Spectrum Cigarette; Other: Low nicotine level e-liquid; Other: Tobacco Flavors
- NNC cigarette + moderate nicotine e-liquid + variety flavors (Experimental): Participants are provided with normal nicotine content tobacco Spectrum Cigarettes along with moderate nicotine level e-liquid cartridges and can choose from tobacco and non-tobacco e-liquid flavors.
  Interventions: Other: NNC Spectrum Cigarette; Other: Moderate nicotine level e-liquid; Other: Tobacco and non-tobacco e-liquid flavors
- NNC cigarette + low nicotine e-liquid + variety flavors (Experimental): Participants are provided with normal nicotine content tobacco Spectrum Cigarettes along with very low or nicotine-free nicotine level e-liquid cartridges and can choose from tobacco and non-tobacco e-liquid flavors
  Interventions: Other: NNC Spectrum Cigarette; Other: Low nicotine level e-liquid; Other: Tobacco and non-tobacco e-liquid flavors
- Very Low Nicotine Content (VLNC) cigarette + moderate nicotine e-liquid + tobacco flavor (Experimental): Participants are provided with very low nicotine content tobacco Spectrum Cigarettes along with moderate nicotine level e-liquid cartridges and can choose from tobacco e-liquid flavors.
  Interventions: Other: VLNC Spectrum Cigarette; Other: Moderate nicotine level e-liquid; Other: Tobacco Flavors
- VLNC cigarette + low nicotine e-liquid +tobacco flavors (Experimental): Participants are provided with very low nicotine content tobacco Spectrum Cigarettes along with very low or nicotine-free nicotine level e-liquid cartridges and can choose from tobacco e-liquid flavors.
  Interventions: Other: VLNC Spectrum Cigarette; Other: Low nicotine level e-liquid; Other: Tobacco Flavors
- VLNC cigarette + moderate nicotine e-liquid + variety flavors (Experimental): Participants are provided with very low nicotine content tobacco Spectrum Cigarettes along with moderate nicotine level e-liquid cartridges and can choose from tobacco and non-tobacco e-liquid flavors.
  Interventions: Other: VLNC Spectrum Cigarette; Other: Moderate nicotine level e-liquid; Other: Tobacco and non-tobacco e-liquid flavors
- VLNC cigarette + low nicotine e-liquid + variety flavors (Experimental): Participants are provided with very low or nicotine-free nicotine content tobacco Spectrum Cigarettes along with very low nicotine level e-liquid cartridges and can choose from tobacco and non-tobacco e-liquid flavors
  Interventions: Other: VLNC Spectrum Cigarette; Other: Low nicotine level e-liquid; Other: Tobacco and non-tobacco e-liquid flavors

INTERVENTIONS:
Other: NNC Spectrum Cigarette — Participants are provided with normal nicotine content Spectrum Cigarette for 13 weeks.
  Arms: NNC cigarette + low nicotine e-liquid + tobacco flavors; NNC cigarette + low nicotine e-liquid + variety flavors; NNC cigarette + moderate nicotine e-liquid + variety flavors; Normal Nicotine Content (NNC) cigarette + moderate nicotine e-liquid + tobacco flavors
Other: VLNC Spectrum Cigarette — Participants are provided with very low nicotine content Spectrum Cigarette for13 weeks
  Arms: VLNC cigarette + low nicotine e-liquid + variety flavors; VLNC cigarette + low nicotine e-liquid +tobacco flavors; VLNC cigarette + moderate nicotine e-liquid + variety flavors; Very Low Nicotine Content (VLNC) cigarette + moderate nicotine e-liquid + tobacco flavor
Other: Moderate nicotine level e-liquid — Participants are provided with moderate nicotine level e-liquid for 13 weeks
  Arms: NNC cigarette + moderate nicotine e-liquid + variety flavors; Normal Nicotine Content (NNC) cigarette + moderate nicotine e-liquid + tobacco flavors; VLNC cigarette + moderate nicotine e-liquid + variety flavors; Very Low Nicotine Content (VLNC) cigarette + moderate nicotine e-liquid + tobacco flavor
Other: Low nicotine level e-liquid — Participants are provided with very low or nicotine-free nicotine level e-liquid for 13 weeks
  Arms: NNC cigarette + low nicotine e-liquid + tobacco flavors; NNC cigarette + low nicotine e-liquid + variety flavors; VLNC cigarette + low nicotine e-liquid + variety flavors; VLNC cigarette + low nicotine e-liquid +tobacco flavors
Other: Tobacco Flavors — Participants can choose e-liquid flavors from a selection of tobacco flavors
  Arms: NNC cigarette + low nicotine e-liquid + tobacco flavors; Normal Nicotine Content (NNC) cigarette + moderate nicotine e-liquid + tobacco flavors; VLNC cigarette + low nicotine e-liquid +tobacco flavors; Very Low Nicotine Content (VLNC) cigarette + moderate nicotine e-liquid + tobacco flavor
Other: Tobacco and non-tobacco e-liquid flavors — Participants can choose e-liquid flavors from a selection of flavors that includes tobacco and non-tobacco choices
  Arms: NNC cigarette + low nicotine e-liquid + variety flavors; NNC cigarette + moderate nicotine e-liquid + variety flavors; VLNC cigarette + low nicotine e-liquid + variety flavors; VLNC cigarette + moderate nicotine e-liquid + variety flavors

SUMMARY:
Project 2 will evaluate the impact of very low nicotine content cigarettes, e-cigarette nicotine content, and e-cigarette flavoring on cigarettes smoked per day, nicotine exposure, puff topography, discomfort/dysfunction, other health-related behaviors, nicotine/tobacco dependence, biomarkers of tobacco exposure, intention to quit, compensatory smoking, other tobacco use, cardiovascular function, and perceived risk. Project 2 will also evaluate differences between conditions in compliance with product use and the ability to abstain from cigarette smoking when provided a financial incentive for abstinence from combusted tobacco. This is not a treatment program for smoking.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who have tried vaping multiple times.
* Generally good health.

Exclusion Criteria:

* If female, currently pregnant, trying to become pregnant or breastfeeding.
* Planning to quit smoking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Donny, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Wake Forest Biotech Place, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to other researchers, please contact the principal investigator for instructions.

REFERENCES:
- [Background] Agaku IT, King BA, Husten CG, Bunnell R, Ambrose BK, Hu SS, Holder-Hayes E, Day HR; Centers for Disease Control and Prevention (CDC). Tobacco product use among adults--United States, 2012-2013. MMWR Morb Mortal Wkly Rep. 2014 Jun 27;63(25):542-7. PMID 24964880
- [Background] Arrazola RA, Singh T, Corey CG, Husten CG, Neff LJ, Apelberg BJ, Bunnell RE, Choiniere CJ, King BA, Cox S, McAfee T, Caraballo RS; Centers for Disease Control and Prevention (CDC). Tobacco use among middle and high school students - United States, 2011-2014. MMWR Morb Mortal Wkly Rep. 2015 Apr 17;64(14):381-5. PMID 25879896
- [Background] Baker H. E-cigarettes and subsequent tobacco use in adolescence. Lancet Oncol. 2015 Oct;16(13):e481. doi: 10.1016/S1470-2045(15)00272-7. Epub 2015 Aug 28. No abstract available. PMID 26321209
- [Background] Bandiera FC, Ross KC, Taghavi S, Delucchi K, Tyndale RF, Benowitz NL. Nicotine Dependence, Nicotine Metabolism, and the Extent of Compensation in Response to Reduced Nicotine Content Cigarettes. Nicotine Tob Res. 2015 Sep;17(9):1167-72. doi: 10.1093/ntr/ntu337. Epub 2015 Jan 2. PMID 25555385
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Biener L, Abrams DB. The Contemplation Ladder: validation of a measure of readiness to consider smoking cessation. Health Psychol. 1991;10(5):360-5. doi: 10.1037//0278-6133.10.5.360. PMID 1935872
- [Background] Benowitz NL, Pomerleau OF, Pomerleau CS, Jacob P 3rd. Nicotine metabolite ratio as a predictor of cigarette consumption. Nicotine Tob Res. 2003 Oct;5(5):621-4. doi: 10.1080/1462220031000158717. PMID 14577978
- [Background] Benowitz NL, Henningfield JE. Establishing a nicotine threshold for addiction. The implications for tobacco regulation. N Engl J Med. 1994 Jul 14;331(2):123-5. doi: 10.1056/NEJM199407143310212. No abstract available. PMID 7818638
- [Background] Benowitz NL, Dains KM, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P 3rd. Progressive commercial cigarette yield reduction: biochemical exposure and behavioral assessment. Cancer Epidemiol Biomarkers Prev. 2009 Mar;18(3):876-83. doi: 10.1158/1055-9965.EPI-08-0731. Epub 2009 Mar 3. PMID 19258480
- [Background] Benowitz NL, Dains KM, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P 3rd. Smoking behavior and exposure to tobacco toxicants during 6 months of smoking progressively reduced nicotine content cigarettes. Cancer Epidemiol Biomarkers Prev. 2012 May;21(5):761-9. doi: 10.1158/1055-9965.EPI-11-0644. Epub 2012 Feb 21. PMID 22354905
- [Background] Benowitz NL, Hall SM, Stewart S, Wilson M, Dempsey D, Jacob P 3rd. Nicotine and carcinogen exposure with smoking of progressively reduced nicotine content cigarette. Cancer Epidemiol Biomarkers Prev. 2007 Nov;16(11):2479-85. doi: 10.1158/1055-9965.EPI-07-0393. PMID 18006940
- [Background] Benowitz NL, Nardone N, Dains KM, Hall SM, Stewart S, Dempsey D, Jacob P 3rd. Effect of reducing the nicotine content of cigarettes on cigarette smoking behavior and tobacco smoke toxicant exposure: 2-year follow up. Addiction. 2015 Oct;110(10):1667-75. doi: 10.1111/add.12978. Epub 2015 Jul 21. PMID 26198394
- [Background] Blank MD, Disharoon S, Eissenberg T. Comparison of methods for measurement of smoking behavior: mouthpiece-based computerized devices versus direct observation. Nicotine Tob Res. 2009 Jul;11(7):896-903. doi: 10.1093/ntr/ntp083. Epub 2009 Jun 11. PMID 19525207
- [Background] Brauer LH, Hatsukami D, Hanson K, Shiffman S. Smoking topography in tobacco chippers and dependent smokers. Addict Behav. 1996 Mar-Apr;21(2):233-8. doi: 10.1016/0306-4603(95)00054-2. PMID 8730526
- [Background] Buchhalter AR, Acosta MC, Evans SE, Breland AB, Eissenberg T. Tobacco abstinence symptom suppression: the role played by the smoking-related stimuli that are delivered by denicotinized cigarettes. Addiction. 2005 Apr;100(4):550-9. doi: 10.1111/j.1360-0443.2005.01030.x. PMID 15784070
- [Background] Butschky MF, Bailey D, Henningfield JE, Pickworth WB. Smoking without nicotine delivery decreases withdrawal in 12-hour abstinent smokers. Pharmacol Biochem Behav. 1995 Jan;50(1):91-6. doi: 10.1016/0091-3057(94)00269-o. PMID 7700960
- [Background] Caggiula AR, Donny EC, White AR, Chaudhri N, Booth S, Gharib MA, Hoffman A, Perkins KA, Sved AF. Cue dependency of nicotine self-administration and smoking. Pharmacol Biochem Behav. 2001 Dec;70(4):515-30. doi: 10.1016/s0091-3057(01)00676-1. PMID 11796151
- [Background] Centers for Disease Control and Prevention (CDC). Cigarette smoking among adults--United States, 2000. MMWR Morb Mortal Wkly Rep. 2002 Jul 26;51(29):642-5. PMID 12186222
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Congress (2009). Family Smoking Prevention and Tobacco Control Act. (H.R. 1256). U. S. Congress. Washington, D.C., U.S. Government Printing Office.
- [Background] Conklin CA, Tiffany ST. Applying extinction research and theory to cue-exposure addiction treatments. Addiction. 2002 Feb;97(2):155-67. doi: 10.1046/j.1360-0443.2002.00014.x. PMID 11860387
- [Background] Cox LS, Tiffany ST, Christen AG. Evaluation of the brief questionnaire of smoking urges (QSU-brief) in laboratory and clinical settings. Nicotine Tob Res. 2001 Feb;3(1):7-16. doi: 10.1080/14622200020032051. PMID 11260806
- [Background] Dawkins L, Turner J, Crowe E. Nicotine derived from the electronic cigarette improves time-based prospective memory in abstinent smokers. Psychopharmacology (Berl). 2013 Jun;227(3):377-84. doi: 10.1007/s00213-013-2983-2. Epub 2013 Jan 24. PMID 23344557
- [Background] Dawkins L, Turner J, Hasna S, Soar K. The electronic-cigarette: effects on desire to smoke, withdrawal symptoms and cognition. Addict Behav. 2012 Aug;37(8):970-3. doi: 10.1016/j.addbeh.2012.03.004. Epub 2012 Mar 10. PMID 22503574
- [Background] Food and Drug Administration, HHS. Deeming Tobacco Products To Be Subject to the Federal Food, Drug, and Cosmetic Act, as Amended by the Family Smoking Prevention and Tobacco Control Act; Restrictions on the Sale and Distribution of Tobacco Products and Required Warning Statements for Tobacco Products. Final rule. Fed Regist. 2016 May 10;81(90):28973-9106. PMID 27192730
- [Background] Dempsey D, Tutka P, Jacob P 3rd, Allen F, Schoedel K, Tyndale RF, Benowitz NL. Nicotine metabolite ratio as an index of cytochrome P450 2A6 metabolic activity. Clin Pharmacol Ther. 2004 Jul;76(1):64-72. doi: 10.1016/j.clpt.2004.02.011. PMID 15229465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 106 screen failures.
Period: Baseline Through Week 12
Arm/Group | Normal Nicotine Content (NNC) Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | Very Low Nicotine Content (VLNC) Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors
Started | 6 | 10 | 5 | 5 | 6 | 6 | 7 | 5
Completed | 2 | 7 | 4 | 4 | 5 | 4 | 4 | 2
Not Completed | 4 | 3 | 1 | 1 | 1 | 2 | 3 | 3
Period: Week 12 Through Day 30 Follow up
Arm/Group | Normal Nicotine Content (NNC) Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | Very Low Nicotine Content (VLNC) Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors
Started | 2 | 7 | 4 | 4 | 5 | 4 | 4 | 2
Completed | 2 | 7 | 4 | 3 | 5 | 4 | 3 | 2
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors: Participants are provided with normal nicotine content tobacco Spectrum Cigarettes along with moderate nicotine level e-liquid cartridges and can choose from tobacco e-liquid flavors.
  NNC Spectrum Cigarette: Participants are provided with normal nicotine content Spectrum Cigarette for 13 weeks.
  Moderate nicotine level e-liquid: Participants are provided with moderate nicotine level e-liquid for 13 weeks
  Tobacco Flavors: Participants can choose e-liquid flavors from a selection of tobacco flavors
- VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor: Participants are provided with very low nicotine content tobacco Spectrum Cigarettes along with moderate nicotine level e-liquid cartridges and can choose from tobacco e-liquid flavors.
  VLNC Spectrum Cigarette: Participants are provided with very low nicotine content Spectrum Cigarette for13 weeks
  Moderate nicotine level e-liquid: Participants are provided with moderate nicotine level e-liquid for 13 weeks
  Tobacco Flavors: Participants can choose e-liquid flavors from a selection of tobacco flavors
- Total: Total of all reporting groups
Arm/Group | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 5 | 5 | 10 | 5 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (7.7) | 43.1 (13.8) | 45.2 (14.4) | 37.8 (11.7) | 42.8 (15.9) | 38 (7.0) | 40.5 (13.3) | 43.8 (11.1) | 41.6 (11.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 4 | 4 | 0 | 2 | 2 | 20
  Male | 3 | 4 | 4 | 2 | 1 | 5 | 7 | 3 | 29
  Prefer not to answer | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 6 | 7 | 6 | 4 | 4 | 4 | 10 | 5 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 4 | 4 | 5 | 2 | 7 | 1 | 30
  Black | 3 | 0 | 2 | 0 | 0 | 2 | 2 | 4 | 13
  More than One Race | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 4
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown/Prefer Not to Answer | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 6 | 6 | 5 | 5 | 10 | 5 | 50

OUTCOME MEASURES:

1. Primary Outcome: Total Cigarettes Smoked Per Day
Description: The average number of cigarettes (study and non-study, summed) smoked per day between the Week 10 and Week 12 visits (the end of the study).
Time Frame: Week 10 through Week 12
Measure: Mean (Standard Deviation); unit: number of cigarettes
Arm/Group | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors
Number analyzed (Participants) | 2 | 4 | 4 | 5 | 4 | 4 | 7 | 2
number of cigarettes | 21.6 (3.7) | 7.7 (12.1) | 18.4 (8) | 12.5 (16.3) | 34 (14.8) | 18.7 (13.9) | 17.7 (8.5) | 15.8 (1.1)

2. Secondary Outcome: Measure of Cigarette Exposure Using Expired Carbon Monoxide (CO)
Description: Measure of cigarette smoke exposure using data on expired breath CO. CO was captured using Covita Smokelyzer devices and standard exhalation procedures. The unit of measurement is parts per million (ppm).
Time Frame: Baseline - Week 12
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors
Number analyzed (Participants) | 2 | 4 | 4 | 5 | 4 | 4 | 7 | 2
parts per million (ppm) | 31 (19.8) | 7.2 (3.8) | 18 (7.4) | 12 (7) | 18.2 (3.4) | 21 (7.8) | 18.3 (7.7) | 32.5 (21.9)

3. Secondary Outcome: Number of Subjects With Smoke Free Days
Description: Study team generates the smoke free days outcome by counting days where no cigarettes and no other forms of combusted tobacco products are used. Days where participants use no nicotine products and days where participants only vape are "smoke free." Percentage of smoke free days = the number days that participants reported smoking 0 cigarettes (0 study cigarettes and 0 non-study cigarettes) divided by the total number of days between their randomization and Week 12 visits. Due to the distribution of the data, statisticians grouped participants according to whether they had 0 smoke-free days or more than 0 smoke free days during the study.
Time Frame: Baseline-Week 12
Measure: Number; unit: participants
Arm/Group | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors
Number analyzed (Participants) | 2 | 4 | 4 | 5 | 4 | 4 | 7 | 2
participants
  Subjects with 0% smoke free days | 1 | 1 | 3 | 3 | 4 | 3 | 6 | 0
  Subjects with more than 0% smoke free days | 1 | 3 | 1 | 2 | 0 | 1 | 1 | 2

4. Other Pre Specified Outcome: Minnesota Nicotine Withdrawal Scale
Description: Measure of discomfort and dysfunction; 15-item self-reported scale to evaluate the effects of smoking cessation. Score ranges from 0 to 60 with higher score denoting more severe symptoms.
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Days Using Assigned Vaping Device
Description: collected through Interactive Voice Response (IVR) Review
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cigarette Evaluation Scale
Description: Assesses the extent to which the product they just sampled produced various subjective effects including satisfaction, good taste, dizziness, reduced appetite, nausea, and enjoyable sensations in the throat and chest. Score ranges from 1 to 91 with a higher score denoting more positive sensations.
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Mercapturic Acids
Description: Measure of toxicant exposure
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Fagerstrom Nicotine Dependence Scale
Description: Dependence Measure
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Study Cigarettes Smoked Per Day
Description: Study cigarettes smoked per day
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

10. Other Pre Specified Outcome: IVR Review and Timeline Followback and E-liquid Accountability
Description: Measure of vaping device use
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Choices to Smoke in Preference Assessment Task
Description: Measure of relative reinforcement
Time Frame: Week 00
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Purchase Task
Description: Measure of relative reinforcement and substitution
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Predicted Behavior Questionnaire
Description: Measure of hypothetical cigarette and vaping device use
Time Frame: Week 12
Reporting Status: Not Posted

14. Other Pre Specified Outcome: IVR Review and Timeline Followback
Description: Measure of compliance
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Drop-out Rate
Description: Drop-out rate
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Urge to Use Questionnaire
Description: Measure of discomfort and dysfunction
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Center for Epidemiologic Studies Depression Scale
Description: Measure of discomfort and dysfunction
Time Frame: Baseline, Weeks 04, 08, 12
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Breath Alcohol
Description: Alcohol use
Time Frame: Baseline - Week 12
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Urine Drug Screen
Description: Drug use
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Alcohol Use Questionnaire
Description: Alcohol use
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Drug Use Questionnaire
Description: Drug use
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Weight
Description: Weight
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Urinary Anatabine Biomarker
Description: Measure of cigarette exposure and compliance
Time Frame: Baseline -Week 12
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Total Nicotine Equivalents
Description: Measure of nicotine exposure
Time Frame: Baseline - Week 12
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Environmental and Social Influences on Tobacco Use Questionnaire
Description: Measure of smoking and vaping context
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Context of Product Use Questionnaire
Description: Measure of smoking and vaping context
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Puff Topography
Description: Measure of smoking and vaping topography
Time Frame: Weeks 01 and 10
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Vaping Utility Questionnaire
Description: Measure of product expectancy
Time Frame: Baseline, Week 12
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Smoking and Vaping Expectancy Questionnaires
Description: Measure of product expectancy
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Cigarette and Product Evaluation Scale
Description: Measure of product characteristics
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Perceived Health Risk Questionnaire
Description: Measure of perceived personal health risk
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Penn State Smoking Dependence Questionnaire
Description: Dependence Measure (smoking and vaping)
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Primary Subscales From Brief Wisconsin Inventory of Smoking Dependence Motive (WISDM)
Description: Dependence Measure
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Population Assessment of Tobacco and Health (PATH) Smoking Dependence Questions
Description: Dependence Measure (smoking and vaping)
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Stages of Change
Description: Measure of intention to quit
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Contemplation Ladder
Description: Measure of intention to quit
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Quit Attempts
Description: Measure of intention to quit
Time Frame: Baseline-Week 12
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Post-intervention Changes in Tobacco Use Behavior
Description: Measure of 30-day tobacco use post-intervention of study products
Time Frame: 30 Day Follow up
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Qualitative Interview
Description: Themes related to product use patterns, e-liquid flavor selection, non-compliance and general study feedback
Time Frame: 30 Day Follow up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline through 12 weeks
Groups:
- Pre-Randomization: Participants signed consent but screen failed before randomizing into study
Arm/Group | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors | Pre-Randomization
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6 | 0/5 | 0/5 | 0/10 | 0/5 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6 | 0/5 | 1/5 | 1/10 | 0/5 | 0/106
Other Adverse Events (participants affected / at risk) | 4/6 | 6/7 | 6/6 | 6/6 | 5/5 | 4/5 | 10/10 | 4/5 | 14/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors (N=6) | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors (N=7) | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors (N=6) | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor (N=6) | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors (N=5) | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors (N=5) | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors (N=10) | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors (N=5) | Pre-Randomization (N=106)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
anaphylaxis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavors (N=6) | VLNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors (N=7) | VLNC Cigarette + Low Nicotine E-liquid +Tobacco Flavors (N=6) | VLNC Cigarette + Moderate Nicotine E-liquid + Tobacco Flavor (N=6) | NNC Cigarette + Low Nicotine E-liquid + Variety Flavors (N=5) | NNC Cigarette + Moderate Nicotine E-liquid + Variety Flavors (N=5) | NNC Cigarette + Low Nicotine E-liquid + Tobacco Flavors (N=10) | VLNC Cigarette + Low Nicotine E-liquid + Variety Flavors (N=5) | Pre-Randomization (N=106)
Lymph Node, pain (swollen) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (slow heart rate) (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (ache/fullness) (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tingling sensation left ear (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Ache (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (upset stomach) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal Reflux (GERD/heartburn/acid) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth decay (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (frustration) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis - sinus infection (incl. bacterial, fungal, viral) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sprained Ankle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appetite, Increase/hunger (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (low blood sugar) (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (muscle aches/pain/spasms) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Arthralgia (joint aches) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exposed Jaw Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness/Lightheadedness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Headache (incl. migraine) (Vascular disorders) | 1 (3) | 2 (2) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 1 (1)
Intracranial Vascular Event (stroke/aneurysm) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (numbness/tingling) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety, clinical diagnosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxious (nervous) mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety/Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CES-D Score, elevated (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (5) | 3 (3) | 3 (4) | 1 (1) | 6 (6)
Depressed (sad) mood (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (change/disturbance in sleep) (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nightmare/terror (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forgetfulness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Worsened Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (incl. seasonal allergies) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (General disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Cough, Productive (lung 'fullness') (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nasal congestion (incl. runny nose) (General disorders) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 2 (3) | 2 (2) | 2 (3) | 3 (3) | 1 (1)
Nosebleed / Dry nasal membrane (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal Drip (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sore throat (incl. itchy/irritated throat) (Hepatobiliary disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Hyperhidrosis (excessive sweating) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Hypertension (high BP) (Cardiac disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
methicillin-resistant Staphylococcus aureus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cut/Abrasion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
torn hamstring tendon (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
stiffness thumb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
elevated potassium (hyperkalemia) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/46/NCT03185546/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT03185546/ICF_002.pdf